CLINICAL TRIAL: NCT06348030
Title: Totally Robotic Versus Surgeon-Assisted Robotic Lung Resection For Early-Stage Non-Small Cell Lung Cancer: A Randomized Controlled Trial
Brief Title: Totally Robotic Versus Surgeon-Assisted Robotic Lung Resection For Early-Stage NSCLC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Wael Hanna, Division Head & Associate Professor, Division of Thoracic Surgery, McMaster University, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17401
Record Dates: First submitted 2024-03-28; First posted 2024-04-04 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgeon-Assisted (Active Comparator): Patients randomized to this arm will undergo RTS with the Medtronic Signia Stapler.
  Interventions: Device: Medtronic Signia Stapler
- Totally Robotic (Experimental): Patients randomized to this arm will undergo RTS with the Da Vinci Vessel Sealer Extend Energy Device and SureForm Stapler.
  Interventions: Device: Vessel Sealer Extend Energy Device and SureForm Stapler

INTERVENTIONS:
Device: Medtronic Signia Stapler — The Signia Stapler is a powered stapler that can be used for tissue dissection and vessel sealing during surgery.
  Arms: Surgeon-Assisted
Device: Vessel Sealer Extend Energy Device and SureForm Stapler — The Vessel Sealer Extend Energy Device is integrated with the da Vinci system and uses bipolar energy technology to facilitate tissue dissection and vessel sealing.
  Arms: Totally Robotic

SUMMARY:
Robotic-assisted thoracoscopic surgery (RTS) is safe and effective for patients with early-stage non-small cell lung cancer (NSCLC). During RTS, division, dissection, and sealing of lung tissue, bronchi, and blood vessels can be performed using handheld staplers with assistance from a bedside surgeon (Surgeon-Assisted), or totally robotically with robotic staplers and energy devices by the console surgeon (Totally Robotic). Totally Robotic lung resection enables the operating surgeon to perform the case independently, but its implication on costs and patient outcomes remains unknown. There also is, however, a lack of prospective research evaluating the costs of the two methods for dissection and vessel sealing in RTS. This RCT aims to evaluate the costs and perioperative patient outcomes of Totally Robotic lung resection using the Vessel Sealer Extend energy device (for vessels <7mm) and the SureForm robotic stapler (Intervention) versus Surgeon-Assisted robotic lung resection using the Signia stapler (Control) during RTS for NSCLC using the da Vinci system.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 120 years at time of consent
* Ability to speak and understand English
* Clinical stage I, II or IIIa NSCLC
* Candidate for RTS, as determined by the operating surgeon

Exclusion Criteria:

* Anticoagulation with inability to cease anticoagulant therapy prior to surgery
* Incurable coagulopathy
* Systemic vascular disease or vasculitis
* Not a candidate for RTS

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Costs of Totally Robotic versus Surgeon-Assisted Robotic Lung Resection | Up to 3 weeks following hospital discharge
  Surgical device (stapler or energy) costs per surgery, along with inpatient hospitalization costs per day following surgery will be collected and evaluated in Canadian dollars.

SECONDARY OUTCOMES:
Operating Room Time | 3 weeks post-surgery
  Entry into Operating Room to Exit, in minutes
Length of Stay in Hospital | 3 weeks post-surgery
  Admission Date to Discharge Date, in days
Duration of Chest Tube | 3 weeks post-surgery
  Insertion Date to Discharge Date, in days
Intraoperative Complications and Adverse events (AEs) | 3 weeks post-surgery
  Short-term clinical outcomes, as measured by intraoperative complications and postoperative AEs, will be recorded during patient follow-ups.

CONTACTS AND LOCATIONS:
Overall Officials: Waël C Hanna, MDCM, MBA, FRCSC, Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No